CLINICAL TRIAL: NCT00069368
Title: ORWH:SCOR on Sex and Gender Factors Affecting Women's Incontinence
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: ORSCOR dk64538 (completed); P50DK064538 (NIH)
Record Dates: First submitted 2003-09-24; First posted 2003-09-26 (Estimated); Last update posted 2025-05-04 (Actual); Status verified 2014-09

CONDITIONS: Urinary Incontinence; Diabetes
Keywords: Healthy
MeSH Terms: conditions — Urinary Incontinence; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study consists of two studies with overlapping cohorts. One is a follow up epidemiological study of urinary incontinence, the other is a case control study of lower urinary tract dysfunction in women with diabetes.

Study One:

Subjects for the study will be a retrospective cohort of 2100 middle-aged and older women from a large health maintenance organization who have participated in the Reproductive Risk Factor for Incontinence Study at Kaiser (RRISK). The RRISK I study assembled a retrospective cohort of long-term female Kaiser Permanente members to determine the association between specific childbirth events, hysterectomy, hormone use and urinary incontinence later in life. The study also provides descriptive information on urinary incontinence by type, age, ethnicity, severity and age of onset.

Study Two:

Women with diabetes have a 30-70% increased risk of lower urinary tract dysfunction, including lower urinary tract symptoms, urinary incontinence, and ultimately bladder cystopathy. This sudy investigates the natural history, risk factors, and possible mechanisms of lower urinary tract dysfunction and infection among women with type 2 diabetes as compared to women without diabetes.

ELIGIBILITY:
Previous participation in the Reproductive Risk Factors for Incontinence Study at Kaiser.

Ages: 44 Years to 73 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women aged 40-69 on 1/1/99 who have been Kaiser Permanente members since age 18 and have had half or more of their deliveries at Kaiser Permanente or are nulliparous and have diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 2161 (Actual)
Dates: Start 2003-07; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Urinary Outcomes | 1999-2012

CONTACTS AND LOCATIONS:
Overall Officials: Jeanette Brown, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Kaiser Permanente, Northern California, Division of Research, Oakland, California, United States